CLINICAL TRIAL: NCT00206206
Title: Evaluation of an ICU Hyperglycemia Protocol Using Insulin Aspart.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Atlantic Health System (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R05-04-002
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2006-02-07 (Estimated); Status verified 2005-09

CONDITIONS: Hyperglycemia
MeSH Terms: conditions — Hyperglycemia

INTERVENTIONS:
Procedure: Hyperglycemia Protocol Procedure

SUMMARY:
In response to the evidence supporting "tight" glucose control (70 - 110) in the critical care setting, the MMH ICU developed a protocol utilizing regular intravenous insulin. This protocol was initiated in 2002. Monitoring of the data collected revealed effective glycemic control when this protocol was used. However, limited utilization has led to overall ineffective glycemic control in this ICU. The poor utilization is largely due to a general reluctance of physicians to start their patients on an intravenous insulin infusion. As contributing to this poor compliance is the "open" nature of the ICU. The MMH ICU is an "open" ICU, meaning that many physicians across multiple subspecialties admit to this unit. Approaches to controlling hyperglycemia vary greatly, depending largely upon the treating physician. In an attempt to improve overall glycemic control in this "open" ICU, the Subcutaneaous Insulin Aspart Hyperglycemia Protocol (SIAP) was developed which incorporates a subcutaneous insulin aspart regimen that triggers the use of a regular insulin infusion protocol when the SIAP is not adequately controlling the patient's blood glucose.

This study aims to evaluate 1) the effect the SIAP on overall glycemic control in the ICU, 2) the effectiveness that the SIAP has on controlling blood glucose as compared with past practices using regular insulin, and 3) the effect the SIAP has on patient complications and outcomes in the MMH ICU.

ELIGIBILITY:
Inclusion Criteria: Valid physician order of the protocol. -

Exclusion Criteria: No valid phycician order for the protocol

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235
Dates: Start 2005-07

PRIMARY OUTCOMES:
1) to evaluate the effect a subcutaneous insulin aspart hyperglycemia protocol on overall glycemic control in an ICU.
2) to evaluate the effect an insulin aspart hyperglycemia protocol has on controlling blood glucoses as compared with past practices of a regular insulin regimen.
3) to assess the effect a hyperglycemis i9nsulin aspart protocol has on patient outcomes in this ICU

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Griffith, Principal Investigator — Moristown Memorial Hospital
Locations (1):
- Morristown Memorial hospital, Morristown, New Jersey, United States